CLINICAL TRIAL: NCT04067869
Title: Participation of Cytomegalovirus Infection or an Autoimmune Process in T Lymphocyte Activation of HIV-1 Infected Patients With Undetectable Viral Load on Antiretroviral Therapy.
Brief Title: Cytomegalovirus Infection in Patients With HIV-1 Infection
Acronym: ACTHIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2009/22
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cytomegalovirus Infections; HIV-1-infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Patient with confirmed HIV-1 infection
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — Blood sample containing 3 ethylene-diamine-tetra-acetic acid tubes (7ml), 3 dry tubes (7ml) and 5 citrated tubes, ie 9 tubes

SUMMARY:
The purpose of this study is to assess the level of CD4 and CD8 T cell activation in an observational cohort study of HIV-1 patients, virosuppressed on combined antiretroviral therapy (< 50 copies/ml) for at least 2 years and to focus on two factors that could participate in this activation: cytomegalovirus infection and auto-immune disorders.

DETAILED DESCRIPTION:
T cell activation plays a central role in HIV pathogenesis and is highly correlated to disease progression even in HIV patients virosuppressed on combined antiretroviral therapy since years. The mechanisms underlying this activation in virosuppressed patients are poorly understood. Identifying some factors involved in immune activation that can be targeted by therapies could optimize the treatment of HIV patients. The purpose of this study is to assess the level of CD4 and CD8 T cell activation in an observational cohort study of HIV-1 patients, virosuppressed on combined antiretroviral therapy (< 50 copies/ml) for at least 2 years and to focus on two factors that could participate in this activation: cytomégalovirus infection and auto-immune disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the Aquitaine ANRS CO3 cohort aged 18 years or older (confirmed HIV-1 infection and at least one follow-up in the cohort),
* plasma HIV-1 RNA <50 copies / ml for at least 24 months under a highly active antiretroviral combination (treatment comprising at least 3 antiretroviral drugs) modified or initiated between 2005 and 2008,
* Follow-up in one of the departments of Bordeaux University Hospital or Libourne Hospital,
* Free, informed and written consent, signed by the patient and the investigator (Consent of the Aquitaine CO3 Cohort and linked to this specific study).

Exclusion Criteria:

* Presence of 2 consecutive measurements of HIV RNA> 50 copies / ml,
* History of immunotherapy treatments (interleukin-2),
* Hepatitis B or C co-infections,
* Pregnancy
* Breastfeeding
* Symptomatic infectious episode in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2010-02-16 (Actual); Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-13 (Actual)

PRIMARY OUTCOMES:
Measurement of systemic lymphocyte activation | At the screening
  Measured by the expression of HLA-DR and CD38 markers on the surface of CD4 + and CD8 + LT by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle PELLEGRIN, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No